CLINICAL TRIAL: NCT07128589
Title: Clinical Evaluation of 3M(TM) Filtek(TM) Supreme Flowable Composites for Class IV and Veneers
Brief Title: 3M(TM) Filtek(TM) Supreme Flowable Composites for Class IV and Veneers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-00581
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Dental Restoration; Dental Veneers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Class IV Restoration (Experimental): 3MTM FiltekTM Supreme Flowable Composites in class IV restoration
  Interventions: Device: 3MTM FiltekTM Supreme Flowable Composite
- Veneers (Experimental): 3MTM FiltekTM Supreme Flowable Composites in veneers
  Interventions: Device: 3MTM FiltekTM Supreme Flowable Composite

INTERVENTIONS:
Device: 3MTM FiltekTM Supreme Flowable Composite — 3M ™ Supreme Flowable Restorative contains BisGMA,TEGDMA and Procrylat resins. The fillers are a combination of ytterbium trifluoride filler with a range of particles sizes from 0.1 to 5.0 microns, a non-agglomerated/non-aggregated surface modified 20nm silica filler, a non-agglomerated/non/aggregated surface modified 75nm silica filler, and a surface modified aggregated zirconia/silica cluster filler (comprised of 20 nm silica and 4 to 11nm zirconia particles). The aggregate has an average cluster particle size of 0.6 to 10 microns. The inorganic filler loading is approximately 65% by weight (46% by volume).
  3M (TM) Filtek(TM) Supreme Flowable Restorative is a modification of predicate device 3M(TM) Filtek(TM) XT Flowable Restorative (which was a modification of 3M(TM) Filtek(TM) Flow. 3M Filtek Supreme Flowable Composites are used per indication and its approved labeling in this study.

SUMMARY:
This clinical study aims to evaluate the clinical performance of 3M™ Filtek™ Supreme Flowable Composite in class IV and veneer indication. Follow-ups of 7 days, 6, 12, and 24 months will be conducted following an Fédération Dentaire Internationale (FDI) modified score (2023). A minimum of 50 Class IV and 25 veneers will be included in the evaluation. Research data and pictures will be provided for each patient pre-op and at 7 days (baseline, 6 months, 12 months and 24 months. Evaluation will be conducted by two calibrated evaluators different from the operator according to FDI clinical criteria.

DETAILED DESCRIPTION:
Resin composites have been used for anterior restorative solutions as they offer a variety of shades and opacities, reproducing the natural structure correctly. This field in dentistry is increasing as an option for past ceramic restorations, making them accessible and affordable for patients.

The conservative aspect of the adhesive resin composite restorations helped increase the indications for this procedure. Cosmetic contour, also named "no-prep" composite veneers, joined the traditional class III, IV, and V cavities as common indications.

Regular paste composites, used in many layers, are the most adequate option as technique treatment.

Different layers, with specific shades and many levels of opacity/translucency, are combined to reproduce the natural characteristics of teeth. This helps control the shape and dimension of the restoration desired. Nevertheless, the time required for a proper restoration with an esthetic outcome and the need for highly trained skills are the drawbacks for most clinicians.

Flowable consistency composites were developed with some goals to be achieved, such as better adaptation to the cavity, especially in posterior teeth. Additional advantages were a more uncomplicated technique and preventing the resin composite from sticking to the instrument. It has been proved to provide a low elastic modulus layer as a resilient liner before the regular consistency composite restoration. For anterior teeth, flowable composites have been used in clinical evaluations for class V cavities with comparative outcomes concerning regular consistency materials.

Previous evaluations were also conducted for classes I and II in the posterior teeth. Newer, highly filled, flowable composites pushed the traditional techniques for a new injectable technique where a silicone transparent index is made in a previous wax-up field. In this way, a very straight way to reproduce the wax-up is used, guiding the exact shape and texture and overcoming the technical limitations of each professional. The need for clinical data on flowable composites using the injectable technique for anterior veneers and class IV is evident.

Clinical evaluation was done with paste composites used in anterior teeth for composite veneers, which showed a survival rate of 93.4% in a two-year evaluation, similar to 95% of ceramic veneers in the same study. Meijering et al. reported an absolute survival rate of 74% (including absolute and relative failures as endpoints. A retrospective study by Mazzeti et al. described an annual failure rate (AFR) of 9.1% for 5 years and 10% for 10 years. Greisnig et al. (2012) described a survival rate of 87.5% for composite veneers in 3 years and a half, using the USPHS modified method.

A survival rate of 92.86% for class IV restorations was reported for a 4-year evaluation of paste composite resin restorations. Demirci et al. (2018) reported a success rate of 86.2% for a composite brand and 89.7% for another, in a 5-year evaluation of class IV restorations. A Kaplan Meier estimate of 9.9 years showed a survival rate of 74.4% for composite resins used in a class IV cavity.

This single-site, non-randomized, clinical study aims to evaluate the clinical performance of 3M™ Filtek™ Supreme Flowable Composite in class IV and veneer indication. Follow-ups of 7 days, 6, 12, and 24 months will follow a Fédération Dentaire Internationale (FDI) modified score used in previous studies. The last version of the modified FDI score was published in 2023, with an update improving the clarity on scoring the composite restorations. This version of the modified FDI score will be applied in our study. Paste composite survival rates reported by literature are the standard of care for the performance of the flowable composite resin used in our study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 -75 years old
* must be willing and able to provide informed consent to participate in the study
* must be available for the required post-operative follow-up study visits
* must be in good general health
* must be in good oral health hygiene (FMPS < 20%)
* have at least 6 anterior maxillary teeth
* Central and lateral incisors with class IV or Veneer indications. Veneers will be performed exclusively with its contralateral teeth (pairs).

Exclusion Criteria:

* Single tooth veneers
* Canines
* Periodontal disease
* Pulpal diseases
* Occlusal dysfunctions (end-to-end bite)
* Lack of occlusal stability
* Missing posterior teeth, affecting the occlusal distribution
* Study tooth, adjacent tooth, or opposing tooth with mobility > grade 2 using the Miller's tooth mobility index
* Systemic or local disorders that contra-indicate the dental procedures needed in this study
* Rampant, uncontrolled caries
* Heavy use of smoking tobacco (1 pack or equivalent a day) or chewing tobacco
* Evidence of xerostomia
* Evidence of severe bruxing or clenching, or in need of Temporomandibular Joint (TMJ) related therapy
* Known allergic reaction and/or sensitivity to research materials being used
* Condition or history of chronic use of anti-inflammatory, analgesic (pain), and/or mind altering drugs for medical (including psychiatric) and pharmacotherapeutic therapies that might alter the perception of pain
* Tooth surface loss (attrition, erosion, abrasion, or abfraction) on study tooth or adjacent teeth that could impact the perception of pain.
* Taking part in a clinical evaluation of any other dental material
* In the opinion of the Investigator, unsuitable for enrollment in the study for reasons other than those specified in the above exclusion criteria
* Pregnant at the time of enrollment or procedure visit (determined by urine pregnancy test).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Survival of treated site over 24 months | 24 months
  Primary site survival will be based off of an Modified FDI criteria score greater or equal to 4.

SECONDARY OUTCOMES:
Esthetic Properties evaluation | 24 months
  Esthetic quality scores measured on an ordinal scale of 1-5.
Functional Properties evaluation | 24 months
  Functional Properties scores measured on an ordinal scale of 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Allen, DDS, Principal Investigator — NYU College of Dentistry
Locations (1):
- NYU College Of Dentistry, New York, New York, United States

REFERENCES:
- [Background] Ricci WA, Fahl N Jr. Nature-mimicking layering with composite resins through a bio-inspired analysis: 25 years of the polychromatic technique. J Esthet Restor Dent. 2023 Jan;35(1):7-18. doi: 10.1111/jerd.13021. Epub 2023 Feb 6. PMID 36744374
- [Background] Pontons-Melo JC, Atzeri G, Collares FM, Hirata R. Cosmetic recontouring for achieving anterior esthetics. Int J Esthet Dent. 2019;14(2):134-146. PMID 31061994
- [Background] Dietschi D. Free-hand composite resin restorations: a key to anterior aesthetics. Pract Periodontics Aesthet Dent. 1995 Sep;7(7):15-25; quiz 27. PMID 9002903
- [Background] Villarroel M, Fahl N, De Sousa AM, De Oliveira OB Jr. Direct esthetic restorations based on translucency and opacity of composite resins. J Esthet Restor Dent. 2011 Apr;23(2):73-87. doi: 10.1111/j.1708-8240.2010.00392.x. Epub 2011 Feb 25. PMID 21477031
- [Background] Hirata R, Kabbach W, de Andrade OS, Bonfante EA, Giannini M, Coelho PG. Bulk Fill Composites: An Anatomic Sculpting Technique. J Esthet Restor Dent. 2015 Nov-Dec;27(6):335-43. doi: 10.1111/jerd.12159. Epub 2015 Jul 14. PMID 26177219
- [Background] Cieplik F, Scholz KJ, Tabenski I, May S, Hiller KA, Schmalz G, Buchalla W, Federlin M. Flowable composites for restoration of non-carious cervical lesions: Results after five years. Dent Mater. 2017 Dec;33(12):e428-e437. doi: 10.1016/j.dental.2017.09.012. Epub 2017 Nov 6. PMID 29102158
- [Background] Zhang H, Wang L, Hua L, Guan R, Hou B. Randomized controlled clinical trial of a highly filled flowable composite in non-carious cervical lesions: 3-year results. Clin Oral Investig. 2021 Oct;25(10):5955-5965. doi: 10.1007/s00784-021-03901-z. Epub 2021 Apr 2. PMID 33797635
- [Background] Endo Hoshino IA, Fraga Briso AL, Bueno Esteves LM, Dos Santos PH, Meira Borghi Frascino S, Fagundes TC. Randomized prospective clinical trial of class II restorations using flowable bulk-fill resin composites: 4-year follow-up. Clin Oral Investig. 2022 Sep;26(9):5697-5710. doi: 10.1007/s00784-022-04526-6. Epub 2022 May 13. PMID 35556174
- [Background] Rocha Gomes Torres C, Rego HM, Perote LC, Santos LF, Kamozaki MB, Gutierrez NC, Di Nicolo R, Borges AB. A split-mouth randomized clinical trial of conventional and heavy flowable composites in class II restorations. J Dent. 2014 Jul;42(7):793-9. doi: 10.1016/j.jdent.2014.04.009. Epub 2014 Apr 25. PMID 24769385
- [Background] Coachman C, De Arbeloa L, Mahn G, Sulaiman TA, Mahn E. An Improved Direct Injection Technique With Flowable Composites. A Digital Workflow Case Report. Oper Dent. 2020 May/Jun;45(3):235-242. doi: 10.2341/18-151-T. Epub 2020 Feb 26. PMID 32101498
- [Background] Ypei Gia NR, Sampaio CS, Higashi C, Sakamoto A Jr, Hirata R. The injectable resin composite restorative technique: A case report. J Esthet Restor Dent. 2021 Apr;33(3):404-414. doi: 10.1111/jerd.12650. Epub 2020 Sep 11. PMID 32918395
- [Background] Imai A, Takamizawa T, Sugimura R, Tsujimoto A, Ishii R, Kawazu M, Saito T, Miyazaki M. Interrelation among the handling, mechanical, and wear properties of the newly developed flowable resin composites. J Mech Behav Biomed Mater. 2019 Jan;89:72-80. doi: 10.1016/j.jmbbm.2018.09.019. Epub 2018 Sep 17. PMID 30265868
- [Background] Elkaffas AA, Alshehri A, Alqahtani AR, Abuelqomsan MA, Deeban YAM, Albaijan RS, Alanazi KK, Almudahi AF. Randomized Clinical Trial on Direct Composite and Indirect Ceramic Laminate Veneers in Multiple Diastema Closure Cases: Two-Year Follow-Up. Materials (Basel). 2024 Jul 16;17(14):3514. doi: 10.3390/ma17143514. PMID 39063806
- [Background] Meijering AC, Creugers NH, Roeters FJ, Mulder J. Survival of three types of veneer restorations in a clinical trial: a 2.5-year interim evaluation. J Dent. 1998 Sep;26(7):563-8. doi: 10.1016/s0300-5712(97)00032-8. PMID 9754744
- [Background] Mazzetti T, Collares K, Rodolfo B, da Rosa Rodolpho PA, van de Sande FH, Cenci MS. 10-year practice-based evaluation of ceramic and direct composite veneers. Dent Mater. 2022 May;38(5):898-906. doi: 10.1016/j.dental.2022.03.007. Epub 2022 Apr 1. PMID 35379471
- [Background] Gresnigt MM, Kalk W, Ozcan M. Randomized controlled split-mouth clinical trial of direct laminate veneers with two micro-hybrid resin composites. J Dent. 2012 Sep;40(9):766-75. doi: 10.1016/j.jdent.2012.05.010. Epub 2012 Jun 2. PMID 22664565
- [Background] Korkut B, Ozcan M. Longevity of Direct Resin Composite Restorations in Maxillary Anterior Crown Fractures: A 4-year Clinical Evaluation. Oper Dent. 2022 Mar 1;47(2):138-148. doi: 10.2341/20-162-C. PMID 35604829
- [Background] Demirci M, Tuncer S, Sancakli HS, Tekce N, Baydemir C. Five-year Clinical Evaluation of a Nanofilled and a Nanohybrid Composite in Class IV Cavities. Oper Dent. 2018 May/Jun;43(3):261-271. doi: 10.2341/16-358-C. Epub 2018 Mar 13. PMID 29533716
- [Background] van Dijken JW, Pallesen U. Fracture frequency and longevity of fractured resin composite, polyacid-modified resin composite, and resin-modified glass ionomer cement class IV restorations: an up to 14 years of follow-up. Clin Oral Investig. 2010 Apr;14(2):217-22. doi: 10.1007/s00784-009-0287-z. Epub 2009 Jun 6. PMID 19504133
- [Background] Korkut B, Turkmen C. Longevity of direct diastema closure and recontouring restorations with resin composites in maxillary anterior teeth: A 4-year clinical evaluation. J Esthet Restor Dent. 2021 Jun;33(4):590-604. doi: 10.1111/jerd.12697. Epub 2020 Dec 23. PMID 33354867
- [Background] Frese C, Schiller P, Staehle HJ, Wolff D. Recontouring teeth and closing diastemas with direct composite buildups: a 5-year follow-up. J Dent. 2013 Nov;41(11):979-85. doi: 10.1016/j.jdent.2013.08.009. Epub 2013 Aug 15. PMID 23954577
- [Background] Hickel R, Mesinger S, Opdam N, Loomans B, Frankenberger R, Cadenaro M, Burgess J, Peschke A, Heintze SD, Kuhnisch J. Revised FDI criteria for evaluating direct and indirect dental restorations-recommendations for its clinical use, interpretation, and reporting. Clin Oral Investig. 2023 Jun;27(6):2573-2592. doi: 10.1007/s00784-022-04814-1. Epub 2022 Dec 12. PMID 36504246